CLINICAL TRIAL: NCT04114266
Title: Prospective Registry for Patients Undergoing Artificial Urinary Sphincter (AUS) Surgery for Female Stress Urinary Incontinence (SUI) Due to Intrinsic Sphincter Deficiency (ISD)
Brief Title: Registry for Patients Undergoing AUS Surgery for Female SUI Due to ISD
Acronym: VENUS
Status: Active, not recruiting | Type: Observational
Sponsor: European Association of Urology Research Foundation (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: EAU-RF 2019-01
Record Dates: First submitted 2019-09-23; First posted 2019-10-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Stress; Lower Urinary Tract Symptoms; Urination Disorders; Urologic Diseases
Keywords: Urologic Surgical Procedure; Female
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Lower Urinary Tract Symptoms; Urination Disorders; Urologic Diseases | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires on Urinary Incontinence-, Sex Function- and Quality of Life (ICIQ-UI-SF, ICIQ-FLUTSsex, ICIQ-LUTSqol, PGI-I) — Artificial Urinary Sphincter Surgery (Robot-assisted, Laparoscopic, Open, or other) for Female Stress Urinary Incontinence due to intrinsic sphincter deficiency is according to standard practice. Patients scheduled for this type of surgery will be asked to participate in this Registry.
  At baseline and follow-up, the patients will be required to fill in Questionnaires, i.e. ICIQ -Urinary Incontinence - Short Form (ICIQ-UI-SF), ICIQ Female Sexual Matters associated with Lower Urinary Tract Symptoms ( ICIQ-FLUTSsex), ICIQ Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol), Patient Global Impression of Improvement-I (PGI-I) which are commonly used in daily practice to assess urinary incontinence, sexual function and quality of life. During the yearly visits, patients will not be required to come for a clinical visit as the questionnaires and a Follow-up form can be completed by post, e-mail or phone call.

SUMMARY:
Prospective collection of pre-defined parameters of AUS Surgery for Female Stress Urinary Incontinence due to Intrinsic Sphincter Deficiency

DETAILED DESCRIPTION:
This will be a prospective non-controlled cohort study evaluating the outcomes of artificial urinary sphincter (AUS) implantation surgery (Robot-assisted, Laparoscopic, Open or other) in female patients. The data collection will be undertaken from multiple centres in Europe. The participation will be by open invitation from the Urologists from the European Society of Female & Functional Urology Section of the European Association of Urology (ESFFU) to all its members along with other surgeons undertaking these procedures. The aim is to recruit a total of 150 patients in 2 years whereafter patients will be followed until the end of Registry which is 5 years after inclusion of the first patient. There will be no restriction on the number of patients enrolled as long as they are consecutive. The aim is to have a long-term collection of the dataset from as many centres as possible.

An initial assessment for the robustness of the data collection and first clinical evaluation of the data collected will be performed after 1 year by a nominated steering committee. Thereafter, the evaluations will be performed after every year until end of Registry.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be Female and aged over 18 years.
* The patient will undergo an initial AUS implantation surgery (Robot-assisted, Laparoscopic, Open or other) for treatment of stress urinary incontinence due to intrinsic sphincter deficiency.
* Participant is willing and able to give informed consent for participation in the Registry
* Patient is able to complete the questionnaires.

Exclusion Criteria:

- Participating center is unable to contribute consecutive patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients undergoing AUS implantation surgery (Robot-assisted, Laparoscopic, Open or other) for treatment of stress urinary incontinence due to intrinsic sphincter deficiency.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Cure rate | Up to 5 years post surgery
  Cure rate is defined as urinary continence with no pads used or use of 1 light security pad.The cure rate after 5 years of study follow up will be calculated together with its 95% Confidence Intervals, for the total patient group as well as for each of the AUS implantation surgery procedures (Robot-assisted, Laparoscopic, Open, or other).

SECONDARY OUTCOMES:
Time being incontinence-free | Up to 5 years post surgery
  Time being incontinence-free which is defined as the interval being continent after surgery to the date of incontinence recurrence
ICIQ-Urinary Incontinence-Short Form Questionnaire (ICIQ-UI-SF) | At each of the evaluation points up to 5 years post surgery
  The ICIQ-UI-SF is a questionnaire evaluating 4 question items (Frequency or urinary incontinence, Amount of leakage, Overall impact of urinary incontinence, Self-diagnostic item) . The score can range from 0 to 25. Mean ICIQ-UI-SF scores will be calculated at the indicated time points and numbers /percentages of patients in the different surgery categories. Also change in ICIQ-UI-SF score compared to baseline will be calculated.
ICIQ-Female Sexual Matters Associated with Lower Urinary Tract Symptoms (ICIQ-FLUTSsex) | At each of the evaluation points up to 5 years post surgery
  The ICIQ-FLUTSsex is a questionnaire evaluating 4 question items (Pain/discomfort because of dry vagina, Impact of urinary symptoms, Pain with sexual intercourse, Urine leakage with sexual intercourse). The score can range from 0 to 54. Mean ICIQ-FLUTSsex scores will be calculated at the indicated time points and numbers /percentages of patients in the different surgery categories. Also change in ICIQ-FLUTSsex compared to baseline will be calculated.
ICIQ- Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol) | At each of the evaluation points up to 5 years post surgery
  The ICIQ-LUTSqol is a questionnaire evaluating 20 question items on quality of life in urinary incontinent patients with particular reference to social effects. The score can range from 19-76 overall score with greater values indicating increased impact on quality of life.
  Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient. Mean ICIQ-LUTSqol scores will be calculated at the indicated time points and numbers /percentages of patients in the different surgery categories. Also change in ICIQ-LUTSqol compared to baseline will be calculated.
24-hour pad tests | At each of the evaluation points up to 5 years post surgery
  The results of the 24-hour pad tests (number of pads, grammes of leakage weight) at each of the evaluation points during follow up. The change of results of the 24-hour pad tests will also be compared with baseline over time.
Urodynamic parameter Volume at leakage | At baseline, week 12 after surgery
  The change of the Volume at leakage (ml) will be compared with baseline.
Urodynamic parameter Detrusor overactivity | At baseline, week 12 after surgery
  The change of Detrusor overactivity (yes/no) will be compared with baseline.
Urodynamic parameter Maximum detrusor pressure during pressure-flow study | At baseline, week 12 after surgery
  The change of Maximum detrusor pressure during pressure-flow study (cm H20) will be compared with baseline.
Urodynamic parameter Detrusor pressure at Max flow during pressure-flow study | At baseline, week 12 after surgery
  The change of Detrusor pressure at Max flow during pressure-flow study (cm H20) will be compared with baseline.
Urodynamic parameter Maximum urinary flow during pressure-flow study | At baseline, week 12 after surgery
  The change of Maximum urinary flow during pressure-flow study (ml/s) will be compared with baseline.
Urodynamic parameter Maximum cystometric capacity | At baseline, week 12 after surgery
  The change of Maximum cystometric capacity (ml) will be compared with baseline.
Urodynamic parameter Retrograde leak point pressure | At baseline, week 12 after surgery
  The change of Retrograde leak point pressure (cm H20) will be compared with baseline.
Main conclusion of Urodynamic investigations | At baseline, week 12 after surgery
  Main conclusion of Urodynamic investigations (Pure stress incontinence, Pure urgency incontinence, Mixed stress, urgency incontinence) will be compared with baseline.mic investigation (Pure stress incontinence, Pure urgency incontinence, Mixed stress, urgency incontinence).The change of Urodynamic parameters will be compared with baseline.
Maximum free urinary flow | At baseline, week 6, week 12 after surgery
  The change in Maximum free urinary flow (ml/s) will be compared to baseline.
Post void Residual Volume | At baseline, week 6, week 12 after surgery
  The change in Post void Residual Volume (ml) will be compared to baseline.
Number of patients with complications | During surgery and up to 5 years after surgery
  Type of complications, associated symptoms and whether or not a revision was needed will be recorded.
Time being revision-free | Up to 5 years post-surgery
  The interval from the date of surgery to the date of revision whereby revision is defined as any urogenital surgical intervention that is related to the function, placement, or site reaction to the implanted device
Revision-free rate | At 1, 2, 3, 4, 5 years of Registry follow-up
  The number of patients who are revision-free compared to the total number of patients, whereby revision is defined as any urogenital surgical intervention that is related to the function, placement, or site reaction to the implanted device

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Peyronnet, Dr., Principal Investigator — Rennes University Hospital
Locations (19):
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospital Leuven, Leuven
- Thomayer Hospital, Prague, Czechia
- France (11):
  - University Hospital Bordeaux, Bordeaux
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - Hôpital Lyon Sud, Lyon
  - Hôpital la Conception, Marseille
  - Clinique urologique CHU de NANTES, Nantes
  - University Hospital of Nimes, Nîmes
  - Hôpital de la Pitié-Salpêtrière, Paris
  - University of Rennes, Department of Urology, Rennes
  - CHU Rangueil, Toulouse
  - CHU Nancy, Vandœuvre-lès-Nancy
- Klinikum Lippe, Detmold, Germany
- Maastricht UMC+, Maastricht, Netherlands
- Spain (2):
  - Hospital de La Princesa, Madrid
  - Marqués de Valdecilla University Hospital, Santander
- Addenbrooks Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may share pseudonymised individual data with residents/urologist interested to analyze and publish the results of the registry

REFERENCES:
- See also: EAU Research Foundation Website — https://uroweb.org/eau-research-foundation-eau-rf